CLINICAL TRIAL: NCT04848727
Title: Detection of Atelectasis or Pneumothorax and Resolution With Electrical Impedance Tomography (EIT) in Newborn Infants
Acronym: DePIcT
Status: Completed | Type: Observational
Sponsor: Sharp HealthCare (Other)
Responsible Party: Principal Investigator, Anup Katheria, M.D., Director Neonatal Research Institute, Sharp HealthCare
Other Study IDs: DePIct
Record Dates: First submitted 2021-04-09; First posted 2021-04-19 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Atelectasis Neonatal; Pneumothorax and Air Leak
Keywords: Electrical Impedance Tomography
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atelectasis or Pneumothorax: Infants with asymmetric lung disease (i.e. atelectasis or pneumothorax) confirmed by chest radiograph
  Interventions: Other: Detecting asymmetric lung disease like atelectasis or pneumothorax with electrical impedance tomography (EIT)

INTERVENTIONS:
Other: Detecting asymmetric lung disease like atelectasis or pneumothorax with electrical impedance tomography (EIT) — The EIT system will be placed at the subject's bedside to collect EIT measurements: Ventilation distribution%, changes in regional aeration in arbitrary units (AU), dependent and non-dependent silent spaces. A data acquisition cart will also be placed at the subject's bedside to collect hemodynamic and respiratory parameters measurements including: Heart rate (HR), blood pressure (BP), respiratory rate (RR), fraction of inspired oxygen (FiO2), transcutaneous carbon dioxide (TcCO2), and peripheral oxygen saturation (SpO2) via bedside monitoring devices.
  The LuMon belts for neonates are disposable single-patient use belts that are adhesive-free. EIT measurements and data will be collected on each timeperiods (t1 and t2) for approximately 15-30 minutes on invasive or non-invasive ventilatory support.

SUMMARY:
To validate the benefits of recognizing asymmetric lung disease like atelectasis and pneumothorax in neonatal respiratory distress syndrome using electrical impedance tomography

DETAILED DESCRIPTION:
To quantify the changes in regional lung air content associated with the variations of the respiratory support settings, the following approach will be used. The changes in local air content will be determined in the selected EIT region of interest (ROI) in terms of a change in local average lung density and relative impedance change with respect to a reference air content.

* TimePeriod 1 (t1): The reference lung air content will be measured once the asymmetric lung disease is identified on chest x-ray.
* TimePeriod 2 (t2): A post-lung disease EIT measurement will be obtained at 6-24 hours later or immediately after therapy (i.e. chest tube placement or needle decompression).

Eligible infants with confirmed asymmetric lung disease (atelectasis or pneumothorax) by radiographic images requiring no respiratory support or on mechanical support or nCPAP therapy of 5-8 cm H20 achieved with a ventilator, an underwater "bubble" system, or a variable-flow device will be enrolled. All of these methods of providing the therapy are done with FDA approved devices currently used in the NICU.

EIT data will be acquired using The LuMon Monitor-Neo, GUI software 1.0.x.x/TIC software 1.6.x.xxx (SenTec, Landquart, Switzerland). The EIT system will be placed at the subject's bedside to collect EIT measurements: Ventilation distribution%, changes in regional aeration in arbitrary units (AU), dependent and non-dependent silent spaces.

A data acquisition cart will also be placed at the subject's bedside to collect hemodynamic and respiratory parameters measurements including: Heart rate (HR), blood pressure (BP), respiratory rate (RR), fraction of inspired oxygen (FiO2), transcutaneous carbon dioxide (TcCO2), and peripheral oxygen saturation (SpO2) via bedside monitoring devices.

The LuMon belts for neonates are disposable single-patient use belts that are adhesive-free and consists of 32 electrodes which are sized to the infant's chest circumference, generally at the 4th - 6th rib. Warmed NeoContactAgent (ingredients: Aqua, Glycerol, Sodium chloride) will be applied to the belt before placing on the infant. The embedded position sensor permits the LuMon System to measure and display the patient's position. The soft and expandable closure band prevents the chest from being constrained by the belt and, consequently, prevents restrictions to breathing and increased work of breathing.

EIT measurements and data will be collected on each timeperiods (t1 and t2) for approximately 15-30 minutes on invasive or non-invasive ventilatory support.

The EIT measurements may be repeated on an eligible participant if a reoccurrence of a confirmed asymmetric lung disease, atelectasis or pneumothorax, is identified on a radiographic image.

EIT is currently not used for patient care management at SMBHWN. EIT's use for patient care management is purely experimental. EIT, when used solely for physiologic data collection, its use is not subject to 21 CFR 50, 21 CFR 56, or 21 CFR 812. Data collection via EIT will occur when the subject is in a quiet, sleeping state, and can be accomplished in a convenient time period when care givers or parents are not interacting with the subject.

ELIGIBILITY:
Inclusion Criteria:

1. All infants admitted to the NICU at SMBHWN
2. Informed consent obtained
3. Atelectasis confirmed on CXR
4. Pneumothorax confirmed on CXR

Exclusion Criteria:

1. Declined consent
2. Infants with known congenital anomalies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All infants admitted to the Neonatal Intensive Care Unit (NICU) at Sharp Mary Birch Hospital for Women & Newborns with confirmed asymmetric lung disease (atelectasis or pneumothorax) by radiographic images requiring no respiratory support or on mechanical support or nCPAP therapy of 5-8 cm H20 achieved with a ventilator, an underwater "bubble" system, or a variable-flow device will be enrolled
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2021-08-06 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

PRIMARY OUTCOMES:
Atelectasis: Change in measured % Unventilated Lung between TimePeriods (t1 and t2) | Baseline, pre-intervention/procedure/surgery and Immediately after the intervention/procedure/surgery
  Atelectasis will be calculated using the percentage of the lung fields that are not engaged in tidal volume.(VT)
Pneumothorax: Change in measured % Unventilated Lung between TimePeriods (t1 and t2) | Baseline, pre-intervention/procedure/surgery and Immediately after the intervention/procedure/surgery
  To determine pneumothorax is the percentage of lung areas with non-negligible impedance change during breathing.

SECONDARY OUTCOMES:
Geometric Center of Ventilation (CoV) | Baseline, pre-intervention/procedure/surgery and Immediately after the intervention/procedure/surgery
  In the human lung the ideal non-dependent to dependent CoV is 63%. Thus a value of 55% would indicate greater ventilation in the non-dependent lung.
Change in % of total tidal volume (VT) within 8 lung regions | Baseline, pre-intervention/procedure/surgery and Immediately after the intervention/procedure/surgery
  % of total tidal volume will be determined from the trough and peak-to-peak height of the time-volume EIT within the 8 regions of interest
Relative change in uncalibrated aeration (end-expiratory lung volume) | Baseline, pre-intervention/procedure/surgery and Immediately after the intervention/procedure/surgery
  End-expiratory lung volume will be analyzed using four ventral to dorsal regions of interest (ROI) by EIT
Regional distribution of tidal volume | Baseline, pre-intervention/procedure/surgery and Immediately after the intervention/procedure/surgery
  Regional distribution of tidal volume will be analyzed using four ventral to dorsal regions of interest (ROI) by EIT

OTHER OUTCOMES:
Compare respiratory rate | Baseline, pre-intervention/procedure/surgery and Immediately after the intervention/procedure/surgery
  Compare the respiratory rate shown on the LuMon monitor and the one shown on other devices
Compare total impedance from the ventilator and the LuMon device | Baseline, pre-intervention/procedure/surgery and Immediately after the intervention/procedure/surgery
  Compare total impedance from the ventilator and the LuMon device
Compare total volumes from the ventilator and the LuMon Device | Baseline, pre-intervention/procedure/surgery and Immediately after the intervention/procedure/surgery
  Compare total volumes from the ventilator and the LuMon Device

CONTACTS AND LOCATIONS:
Overall Officials: Anup C Katheria, MD, Principal Investigator — Sharp HealthCare
Locations (1):
- Sharp Mary Birch Hospital for Women & Newborns, San Diego, California, United States

REFERENCES:
- [Background] Costa EL, Borges JB, Melo A, Suarez-Sipmann F, Toufen C Jr, Bohm SH, Amato MB. Bedside estimation of recruitable alveolar collapse and hyperdistension by electrical impedance tomography. Intensive Care Med. 2009 Jun;35(6):1132-7. doi: 10.1007/s00134-009-1447-y. Epub 2009 Mar 3. PMID 19255741
- [Background] Miedema M, McCall KE, Perkins EJ, Sourial M, Bohm SH, Waldmann A, van Kaam AH, Tingay DG. First Real-Time Visualization of a Spontaneous Pneumothorax Developing in a Preterm Lamb Using Electrical Impedance Tomography. Am J Respir Crit Care Med. 2016 Jul 1;194(1):116-8. doi: 10.1164/rccm.201602-0292LE. No abstract available. PMID 27367888
- [Background] Rahtu M, Frerichs I, Waldmann AD, Strodthoff C, Becher T, Bayford R, Kallio M. Early Recognition of Pneumothorax in Neonatal Respiratory Distress Syndrome with Electrical Impedance Tomography. Am J Respir Crit Care Med. 2019 Oct 15;200(8):1060-1061. doi: 10.1164/rccm.201810-1999IM. No abstract available. PMID 31091957
- [Background] Kallio M, Rahtu M, van Kaam AH, Bayford R, Rimensberger PC, Frerichs I. Electrical impedance tomography reveals pathophysiology of neonatal pneumothorax during NAVA. Clin Case Rep. 2020 May 24;8(8):1574-1578. doi: 10.1002/ccr3.2944. eCollection 2020 Aug. PMID 32884798
- See also: Design/patents related to the Lumon System — http://www.sentec.com/education/eit/plpm-eit